CLINICAL TRIAL: NCT03664258
Title: Evaluation of the Xpert® Bladder Cancer Monitor Assay Compared to Cystoscopy for the Follow-up of Patients With History of Low or Intermediate Risk Non-muscle-invasive Bladder Cancer (NMIBC): an Observational Prospective International Multicenter Study
Brief Title: A Multi-National Study In Bladder Cancer Patients to Detect Recurrences After TURB (Trans-urethral Resection of the Bladder) Earlier With the Xpert Bladder Cancer Monitor Assay (ANTICIPATE X)
Acronym: ANTICIPATE X
Status: Completed | Type: Observational
Sponsor: Cepheid (Industry)
Collaborators: Axonal-Biostatem (Industry); Stève Consultants (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANTICIPATE X
Record Dates: First submitted 2018-07-25; First posted 2018-09-10 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2021-08

CONDITIONS: Non-muscle-invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Xpert Bladder Cancer Monitor — The Xpert Bladder Cancer Monitor Assay is a qualitative in vitro diagnostic test designed to monitor for the recurrence of bladder cancer in patients previously diagnosed with bladder cancer. It should be used in conjunction with other clinical measures to assess disease recurrence. The test provides a fast and accurate result, is non-invasive and easy to perform.The test utilizes a voided urine specimen and measures the level of five target mRNAs (ABL1, CRH, IGF2, UPK1B, ANXA10) by means of real-time, reverse transcription-polymerase chain reaction (RT-PCR).

SUMMARY:
Bladder cancer is the 5th most common cancer in Europe, with more than 151,000 new cases diagnosed in 2012 (4% of the total). Bladder cancer has the highest recurrence rate of any malignancy, often as high as 70% within 5 years of successful treatment. This high recurrence rate requires diligent and accurate monitoring as a means for early diagnosis and treatment. Considering the burden associated to repeated invasive cystoscopies, there is a need for robust but accurate tests for surveillance. In that prospect, urinary molecular tests have been developed although none were deemed adequate in the European clinical guidelines to replace cystoscopies. The Xpert Bladder Cancer Monitor Assay is a qualitative in vitro diagnostic test designed to monitor for the recurrence of bladder cancer in patients previously diagnosed with this cancer. The test provides a fast and accurate result, is non-invasive and easy to perform. The aim of this study is to assess the non-inferiority of the Xpert Bladder Cancer Monitor assay in detecting recurrences in comparison to cystoscopy in the follow-up of patients with low or intermediate risk non-muscle-invasive bladder cancer (NMIBC).

DETAILED DESCRIPTION:
Patient recruitment and follow-up are closed. The study is in analysis phase.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing a follow-up cystoscopy at the time of enrolment for low or intermediate risk NMIBC patients in the follow-up phase (according to the 2017 EAU guidelines),
* Patient must accept to be followed for 1 year after enrolment cystoscopy,
* Patient who can provide urine samples naturally (e.g. no catheterization),
* 18 years or older at the time of enrolment,
* Signed informed consent.

Exclusion Criteria:

* Patient with history of NMIBC stratified at the time of enrolment as high risk according to 2017 EAU Guidelines,
* Patient with history of Muscle-Invasive Bladder Cancer (MIBC),
* Patient having undergone a TURB less than 3 months before enrolment,
* Patient having received Mitomycin C (MMC) or Bacillus Calmette-Guerin (BCG) intravesical instillations less than 3 months before enrolment (a single MMC post-operative instillation is acceptable for inclusion).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with low or intermediate risk NMIBC and included in a monitoring program are considered for the study. Patients are recruited within the medical consultation of the Urology departments of the study sites (hospitals, clinics) and registered following a chronological order.
Sampling Method: Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the comparison of the number of recurrences detected between the standard of care (cystoscopy) and a urine biomarker assay | 12 months from patient enrollment in the study.
  The primary outcome measure is the ratio of patients presenting recurrence, comparing the number of patients with positive cystoscopies over the duration of 12 months to the number of patients with positive Xpert Bladder Cancer Monitor Assay at D0 (at enrollment).

SECONDARY OUTCOMES:
Comparison of the number of patients with negative Xpert Bladder Cancer Monitor assay results and the number of patients with negative cystoscopy results at D0 who are not presenting with recurrent bladder cancer within 12 months of enrolment cystoscopy. | 12 months from patient enrollment in the study.
  The number of patients with negative Xpert Bladder Cancer Monitor assay results will be compared to the number of patients with negative cystoscopy results at D0 who are not presenting with recurrent bladder cancer within 12 months of enrolment cystoscopy. The absence of cancer is defined as absence of suggestion of cancer on cystoscopy performed over 12 months or positive cystoscopy at 12 months not confirmed by TURB.
Comparison of the number of positive and negative tests of Xpert Bladder Cancer Monitor and cystoscopy results at the time of each NMIBC follow-up assessment. | At each patient follow-up up to 12 months of study.
  The number of positive and negative tests of Xpert Bladder Cancer Monitor will be compared to the cystoscopy results at the time of each NMIBC follow-up assessment.
EuroQol Five Dimensions Questionnaire (EQ-5D-5L questionnaire) at Day 0 | At patient enrollment
  Measure of the quality of life of patients with the EQ-5D-5L questionnaire at Day 0 for 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression).
Patient numeric scale for cystoscopy discomfort | At each patient follow-up up to 12 months of study.
  Evaluation of patient's cystoscopy discomfort with a patient numeric scale to complete by the patient after each. The patient self-rates on a 0 (no discomfort) to 10 (maximum discomfort) numeric scale.
Assessment of medical care resources consumption related to bladder cancer at 1 month after each cystoscopy. | 1 month after each cystoscopy through study completion.
  Assessment of medical care resources consumption related to bladder cancer follow-up with the use of a patient questionnaire completed 1 month after each cystoscopy:
  * Number of general practitioner or urologist visits performed during 1 month after the cystoscopy.
  * Number of hospitalization/ duration of hospitalization during 1 month after the cystoscopy
  * Nature of additional medical examination performed during 1 month after the cystoscopy
  * Nature of additional treatments received during 1 month after the cystoscopy
  * Number of sick leave/ duration of sick leave during 1 month after the cystoscopy
EuroQol health visual analogue scale at Day 0. | At patient enrollment.
  Measure of the patient self-rated health on a vertical visual analogue scale numbered from 0 (best health) to 100 (worst health) at Day 0.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Malavaud, M.D., Principal Investigator — CHU Toulouse / Institut Universitaire du Cancer Toulouse Oncopole
Locations (13):
- Austria (2):
  - University Clinic for Urology and Andrology, Salzburg
  - Medical University of Vienna, Vienna
- Teaching Hospital Motol, Prague, Czechia
- CHU Toulouse / Institut Universitaire du Cancer Toulouse Oncopole, Toulouse, France
- Germany (2):
  - Klinikum Braunschweig, Braunschweig
  - University of Regensburg, Regensburg
- Humanitas University - Gradenigo Hospital of Turin, Turin, Italy
- Academic Medical Center, Amsterdam, Netherlands
- Spain (2):
  - Fundacio Puigvert, Barcelona
  - Instituto Valenciano de Oncologia, Valencia
- Sahlgrenska University Hospital, Gothenburg, Sweden
- United Kingdom (2):
  - Royal Surrey County Hospital, Guildford
  - Sunderland City Hospital, Sunderland